CLINICAL TRIAL: NCT05220358
Title: Changes in Immunologic Parameters Following the Addition of Fostemsavir in Virologically Suppressed Immunologic Non-responders Living With HIV-the RECOVER Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Orlando Immunology Center (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OIC_010
Record Dates: First submitted 2022-01-31; First posted 2022-02-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
Keywords: CD4 recovery; immunologic recovery; immunologic non responder
MeSH Terms: interventions — fostemsavir

STUDY DESIGN:
Intervention Model Description: self-controlled case series to evaluate the change in immunologic parameters following the addition of FOS to baseline ARV regimens among virologically suppressed INRs through 48 weeks of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FTR+suppressive regimen (Experimental): addition of fostemsavir 600 mg PO BID to the stable suppressive HIV regimen in immunologic non responders
  Interventions: Drug: Fostemsavir 600 MG [Rukobia]

INTERVENTIONS:
Drug: Fostemsavir 600 MG [Rukobia] — FTR 600 mg PO BID added to daily suppressive HIV regimen

SUMMARY:
The RECOVER study is a self-controlled case series to evaluate whether the addition of Fostemsavir (Rukobia) to a stable HIV regimen in virologically suppressed patients living with HIV who never experience optimal CD4 T-cell count recovery can result in meaningful increases in different immunologic parameters such as CD4 T-cell count, CD4 T-cell percentage and CD4/CD8 ratio

DETAILED DESCRIPTION:
In July 2020 the FDA approved fostemsavir (FTR), a prodrug of its active moiety temsavir which is a first-in class attachment inhibitor to be used in combination with other antiretrovirals (ARVs) to treat HIV infection in patients with multi-class drug resistance who are failing their current ARV regimen [1]. FTR is well-tolerated, dosed orally twice-daily, has no food requirement, no need for renal or hepatic dose adjustment and few drug-drug interactions (DDIs) [1-3]. FDA approval was based on 96-week data from the BRIGHTE study which demonstrated that addition of FTR to an optimized background regimen (OBR) among patients with multi-drug resistance failing their current regimen resulted in 96-week virologic suppression rates of 60% among patients with 1-2 fully active ARV classes remaining at baseline (randomized cohort) and 37% among patients with 0 fully active ARV classes remaining at baseline (non-randomized cohort) [4]. Robust CD4+ T-cell recovery was observed with a mean increase of 90 and 205 cells/mm3 through Weeks 24 and 96 respectively among patients in the randomized cohort [4]. The gain in CD4+ T-cells was however most impressive among the most immunocompromised patients, at Week 96 a mean increase of 240 cells/mm3 was observed among those with baseline CD4+ T-cell counts <20 cells/mm3 and 56% of patients with baseline CD4+ T-cell counts <50 cells/mm3 had achieved a CD4+ T-cell count of ≥200 cells/mm3 [4].

These data have raised questions about whether FTR has the ability to promote CD4+ T-cell recovery independently of HIV viral suppression. This first-in-class attachment inhibitor has a unique mechanism of action, the active moiety temsavir binds directly to viral gp120 preventing HIV-1 from interacting with the host immune cell. This process leaves the CD4+ T-cell untouched and it is hypothesized that temsavir binding to gp120 inhibits gp120-mediated apoptosis of CD4+ T-cells and does not allow for activation of other downstream inflammatory pathways that may contribute to CD4+ T-cell death [2]. Other clinical trials of ARVs used in heavily-treatment experienced populations, including those with ibalizumab, dolutegravir, enfuvirtide, maraviroc and etravirine have not demonstrated the degree of CD4+ T-cell recovery observed in the BRIGHTE study [5-9]. Cumulatively these data suggest that FOS may be of benefit in individuals who experience suboptimal immunologic recovery despite achieving viral suppression also known as immunologic non-responders (INRs).

Since 1997, researchers have struggled to identify agents that can restore CD4+T-cell counts and reduce immune activation and inflammation in virologically suppressed INRs [10]. Despite achieving ARV efficacy, this group continues to be at higher risk of disease progression to AIDS, complications related to opportunistic infections (OIs) and death [10, 11]. Recently, data has also revealed that persistent immune activation and inflammation also contributes to higher rates of non-AIDS related events such as hypertension, hyperlipidemia, hyperglycemia and cardiovascular disease [11]. Multiple strategies to address CD4+ T-cell depletion and persistent immune activation among INRs have been investigated over the years, these include the use of adjunctive maraviroc, immune modulators, statins, sitagliptin, niacin, antivirals, nutritional supplements and growth hormone in combination with ART [10, 12-14]. Unfortunately, none of these has demonstrated consistent efficacy and some studies have even revealed loss of virologic control and the occurrence of serious adverse events (AEs) when adjunct therapies were used [10]. These findings highlight an urgent need to identify novel options as adjunct therapy for CD4+T-cell recovery and to reduce inflammation and immune activation among INRs. An ideal agent for this purpose would be well-tolerated, have few DDIs with ARVs and have a low risk of contributing to virologic failure when combined with ARVs. Based on data from the BRIGHTE study, we hypothesize that FTR would be efficacious at establishing significant immune reconstitution in INRs without compromising virologic efficacy or patient safety.

Here, we propose a self-controlled case series to evaluate the change in immunologic parameters following the addition of FTR to baseline ARV regimens among virologically suppressed INRs through 48 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected men or women
* Aged 18-65
* Stable insurance plan
* Documented plasma HIV-1 RNA < 50 c/mL x 2 within the last year prior to screening
* Must be on a stable ARV regimen for ≥6 months prior to screening
* CD4+T-cell count<350 cells/mm3 while on ARVs for at least 2 years
* Must be willing to add FTR 600 mg twice daily to their current antiretroviral regimen
* Must have attended ≥ 2 clinic visits in the 12 months prior to screening

Exclusion Criteria:

* Newly or recently diagnosed HIV-1 infection defined as HIV-1 infection diagnosed in the prior 6 months
* Active HBV or HCV co-infection
* Unstable liver disease or Child-Pugh C liver disease
* History of autoimmune disease
* History of any malignancy ≤5 years
* History of radiation or cytotoxic chemotherapy
* Use of systemic corticosteroids or other immunomodulatory agents in the last 14 days prior to study entry
* Confirmed QT value > 500 msec at Screening or Day 1 or confirmed QTcF value > 470 msec for women and > 450 msec for men at Screening or Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Mean and median change in CD4+T-cell count | 48 weeks
  mean and median change in CD4+T-cell count after the addition of fostemsavir to baseline ARV regimens in virologically suppressed immunologic non responders using pre-fostemsavir values as controls

SECONDARY OUTCOMES:
Mean and median change in CD4+T-cell count | 24 weeks
  mean and median change in CD4+T-cell count after the addition of fostemsavir to baseline ARV regimens in virologically suppressed immunologic non responders using pre-fostemsavir values as controls
mean and median change in CD4+T-cell count percentage | 24 and 48 weeks
  mean and median change in CD4+ percentage after the addition of fostemsavir to baseline ARV regimens in virologically suppressed immunologic non responders using pre-fostemsavir values as controls
mean and median change in CD4/CD8 ratio | 24 and 48 weeks
  mean and median change in CD4/CD8 ratio after the addition of fostemsavir to baseline ARV regimens in virologically suppressed immunologic non responders using pre-fostemsavir values as controls
Proportion with virologic failure defined as an HIV-1 RNA≥50 c/mL | 24 and 48 weeks
  proportion of patients with HIV-1 RNA ≥50 c/mL after the addition of fostemsavir to baseline ARV regimens in virologically suppressed immunologic non responders using pre-fostemsavir values as controls
Safety and tolerability of fostemsavir | Weeks 24 and 48
  Incidence and severity of AEs and laboratory abnormalities and proportion of subjects who discontinue treatment due to AEs
Change in concomitant medications after adding fostemsavir to the baseline ARV regimen over time | Weeks 24 and 48
  Change in number of concomitant medications after the addition of fostemsavir to the baseline ARV regimen using number of concomitant medications pre-fostemsavir as the comparator
Impact of adding fostemsavir to the baseline ARV regimen on medications needed for OI prophylaxis over time | Weeks 24 and 48
  Change in number of concomitant medications for OI prophylaxis after the addition of fostemsavir to the baseline ARV regimen using number of concomitant medications for OI prophylaxis pre-fostemsavir as the comparator
Impact of adding fostemsavir to the baseline ARV regimen on OI incidence and severity over time | Weeks 24 and 48
  Proportion of patients with an incident OI and Change in the severity of incident OIs (grading using the DAIDS grading table)
Assessment of health related quality of life after the addition of fostemsavir to baseline ARV regimens | Weeks 24 and 48
  Change from Baseline in QOL scores using the WHOQOL-HIV BREF
Assessment of HIV or ART-related symptoms after the addition of fostemsavir to baseline ARV regimen | Weeks 24 and 48
  Change from Baseline in health status score using the HIV-SI (HIV-Symptom Index)
Assessment of treatment satisfaction in subjects who have fostemsavir added to their baseline ARV regimen | Weeks 24 and 48
  Change from baseline in treatment satisfaction using the HIV TSQs questionnaire
Assessment of viral resistance in subjects meeting Virologic Rebound Criteria | Weeks 24 and 48
  Incidence of observed genotypic resistance to ARVs for subjects meeting Virologic Rebound Criteria

OTHER OUTCOMES:
Impact of fostemsavir treatment on inflammatory, cellular functional, and viral reservoir biomarkers in immunologic non responders | Weeks 24 and 48
Identification of biomarkers that may predict CD4 recovery and Immunologic non response | Weeks 24 and 48
Evaluation of gp120 detection and correlation with reservoir and inflammatory biomarkers | Weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte-Paige M Rolle, MD, MPH, Principal Investigator — Orlando Immunology Center
Locations (1):
- Orlando Immunology Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No